CLINICAL TRIAL: NCT00359658
Title: Conversion Study to Optimize Immunosuppressive Regimen by Withdrawal of Steroids, Cyclosporine A Dose Reduction and a Switch to Mycophenolatmofetile for Patients After Heart Transplantation in the Long-Term.
Brief Title: Withdrawal of Steroids, Cyclosporine A Dose Reduction and Switch to Mycophenolatmofetile After Heart Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Dr. med. Chhristoph Bara, Clinic for Cardiothoracic, Transplantation and Vascular Surgery, HannoverMS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KKS-94/2004
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Heart Transplantation
Keywords: Cyclosporine; Glucocorticoids; renal insufficiency, chronic; long-term care
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Prednisone; Mycophenolic Acid; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): prednisolon withdrawal: reduction of maintenance dosage, 0,5 mg of the daily dose every week till withdrawal; Mycophenolatmofetile administration: start doses 250 mg, increase of the daily dose about 250 mg every week till reaching 2 g/daily; Cyclosporin A reduction: 8 weeks after starting prednisolon withdrawal and Mycophenolatmofetile administration reduction of Cyclosporin A trough level till a range from 50 to 90 mg/ml
  Interventions: Drug: prednisolon; Drug: Mycophenolatmofetile; Drug: Cyclosporin A

INTERVENTIONS:
Drug: prednisolon — prednisolon withdrawal: reduction of maintenance dosage, 0,5 mg of the daily dose every week till withdrawal
  Other Names: Decortin; steroid withdrawal
Drug: Mycophenolatmofetile — Mycophenolatmofetile administration: start doses 250 mg, increase of the daily dose about 250 mg every week till reaching 2 g/daily
  Other Names: MMF; Cellcept
Drug: Cyclosporin A — Cyclosporin A reduction: 8 weeks after starting prednisolon withdrawal and Mycophenolatmofetile administration reduction of Cyclosporin A trough level till a range from 50 to 90 ng/ml
  Other Names: Sandimmun optoral

SUMMARY:
The purpose of this study is first to improve or save renal function and second to decrease cardiac risk factors by optimising the immunosuppressive regimen by withdrawing steroids and reducing the Cyclosporine A dose. The concomitant administration of Mycophenolatmofetile, an effective immunosuppressive agent, will minimize the risk of acute rejection episodes.

DETAILED DESCRIPTION:
The decrease of quality of life in patients after heart transplantation in the long-term is determined by an increasing incidence of transplant vasculopathy and by immunosuppression-related side effects. Calcineurin inhibitors are associated with chronic nephrotoxicity, while long-term administration of steroids results in an increased incidence of cardiovascular risk factors (e.g. hypertension, lipometabolic disorders, steroid induced diabetes, adipositas)and therefore, carries the potential of graft disfunction.

ELIGIBILITY:
Inclusion Criteria:

* Current immunosuppressive regimen: Cyclosporine A and corticosteroids for at least six month
* Heart transplantation above 3 years dated back
* Serum creatinine < 3,5 mg/dl (310 µmol/l) and BUN < 150 mg/dl
* Cyclosporine A blood level between 50 and 250 ng/ml during the last 12 month

Exclusion Criteria:

* Carcinoma within the last 3 years
* Acute rejection episodes during the last 6 month
* Infection requiring therapeutic intervention
* Hepatitis B, Hepatitis C or HIV infection
* WBC < 3000/µl, haemoglobin < 9g/dl, platelets < 70.000/µl
* Florid gastrointestinal ulcer
* Haemodialysis within the last 4 weeks before study entry
* Pregnancy / lactation
* Administration of other immunosuppressive agents than prescribed
* Mycophenolatmofetile incompatibility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Renal function evaluated by serum creatinine at month 12 and month 24 | month 12 and month 24

SECONDARY OUTCOMES:
Cardiovascular risk factors at month 12 and month 24 | month 12 and month 24
Acute rejection episodes, gastrointestinal disorders and other adverse events at month 12 and month 24 | month 12 and month 24
Quality of life assessed by the SF36, spiroergometry, concomitant medication at month 12 and month 24 | month 12 and month 24

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Bara, Dr. med., Study Director — Hannover Medical School, Department of Thoracic and Cardiovascular Surgery
Locations (1):
- Hannover Medical School, Department of Thoracic and Cardiovascular Surgery, Hanover, Germany

REFERENCES:
- [Derived] Faulhaber M, Mading I, Malehsa D, Raggi MC, Haverich A, Bara CL. Steroid withdrawal and reduction of cyclosporine A under mycophenolate mofetil after heart transplantation. Int Immunopharmacol. 2013 Apr;15(4):712-7. doi: 10.1016/j.intimp.2013.02.012. Epub 2013 Feb 28. PMID 23454241